CLINICAL TRIAL: NCT00597532
Title: Effect of Soy Supplementation on Cellular Markers in Normal and Cancerous Breast Tissue: A Randomized Placebo Controlled Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 02-062
Record Dates: First submitted 2007-12-26; First posted 2008-01-18 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Soy; Milk; Supplementation; 02-062
MeSH Terms: conditions — Breast Neoplasms | interventions — Milk

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): soy (soy protein supplementation 50 grams/day)
  Interventions: Dietary Supplement: Soy
- 2 (Placebo Comparator): milk protein supplementation 50 grams/day
  Interventions: Dietary Supplement: Milk

INTERVENTIONS:
Dietary Supplement: Soy — soy (soy protein supplementation 50 grams/day)
  Arms: 1
Dietary Supplement: Milk — placebo (milk protein supplementation 50 grams/day)
  Arms: 2

SUMMARY:
To Test Effect of Soy Supplementation on Cellular Markers in Normal and Cancerous Breast Tissue using a Randomized Placebo Controlled Study.

Objectives:

* To determine (by immunohistochemistry) whether specific cellular markers and gene products associated with breast carcinoma can be altered by soy therapy.
* To identify genes that can be altered by soy therapy in normal and neoplastic breast tissues by unbiased gene expression analysis using microarrays.
* To compare specific cellular markers and pathways (immunohistochemistry), and gene expression using microarrays in normal and cancerous breast tissue.

DETAILED DESCRIPTION:
Patient Population:

Pre and post menopausal women with breast cancer diagnosed by core needle biopsy scheduled to undergo breast cancer resection for an invasive carcinoma.

Objectives:

* To determine (by immunohistochemistry) whether specific cellular markers and gene products associated with breast carcinoma can be altered by soy therapy.
* To identify genes that can be altered by soy therapy in normal and neoplastic breast tissues by unbiased gene expression analysis using microarrays.
* To compare specific cellular markers and pathways (immunohistochemistry), and gene expression using microarrays in normal and cancerous breast tissue.

Study Design and Intervention Plan:

* Eligible patients will be consented at the time of visit with MSKCC breast surgeon and randomized to receive soy (soy protein supplementation 50 grams/day), or placebo (milk protein supplementation 50 grams/day) over the period until their surgery.
* The diagnostic biopsy (already available at time of appointment with MSKCC surgeon) will be analyzed by immunohistochemistry for proliferation (Ki67) and apoptosis (TUNEL). Additional immunohistochemistry will include HER2, TP53, cyclin D1, p27, BCL2, ER and PR.
* Excision of the breast carcinoma (lumpectomy or mastectomy) will proceed in standard fashion.
* The post-therapy excision specimen will be processed in a standard fashion. Pathologic features, margin status, and tumor size will be assessed by a light microscopic examination of histological sections. In addition to this routine processing, immunohistochemistry assays for proliferation (Ki67), apoptosis (TUNEL), HER2, TP53, cyclin D1, p27, BCL2, ER, and PR will be performed. For correlative biological studies pathologists will select approximately .5 cubic mm representative sections of the neoplastic tissues and normal adjacent breast tissue, which will be snap frozen for gene expression analysis using microarrays.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Breast mass > .5 cm (determined by mammogram, ultrasound, MRI, or palpable criteria)
* Core biopsy diagnosis of invasive carcinoma of the breast

Exclusion Criteria:

* History of active malignancy within previous two years (except for non-melanoma skin cancer and history of breast cancer).
* Regular soy consumption (consumption of more than 3 serving of soy or soy products/supplements per week)
* Allergy to soy or milk protein

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2002-08; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is comparison of the change in proliferation (Ki67) and apoptosis (TUNEL) in cancerous tissue between the 2 groups. | Conclusion of the study

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Shike, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Shike M, Doane AS, Russo L, Cabal R, Reis-Filho JS, Gerald W, Cody H, Khanin R, Bromberg J, Norton L. The effects of soy supplementation on gene expression in breast cancer: a randomized placebo-controlled study. J Natl Cancer Inst. 2014 Sep 4;106(9):dju189. doi: 10.1093/jnci/dju189. Print 2014 Sep. PMID 25190728
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org